CLINICAL TRIAL: NCT06552078
Title: Activation of Biobank for Association Study Between Environmental and Genetic Factors in Inflammatory, Functional and Neoplastic Bilio-pancreatic Diseases
Brief Title: Activation of Biobank Registry for Bilio-pancreatic Diseases
Acronym: BIO-PANCREAS
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Paolo Giorgio Arcidiacono, MD, Professor, IRCCS San Raffaele
Other Study IDs: BIO-PANCREAS
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pancreatitis; Pancreatic Disease; Non-Neoplastic Pancreatic Disorder; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatitis; Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * peripheral blood;
  * portal blood;
  * saliva;
  * urine;
  * stool;
  * cystic fluid;
  * pancreatic juice;
  * biopsy tissue;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of establishing the biobank is to create a collection of biological material and clinical data, with a prospective and retrospective mold, in order to investigate the role of genetic predisposition in multifactorial bilio-pancreatic diseases, so that an evaluation of the possible association in the pathogenesis of exogenous factors with endogenous factors can be allowed.

Multifactorial diseases are in fact an expression of genetic predisposition upon which one or more environmental stimuli act. Usually the aforementioned factors are not capable individually of triggering disease but, when simultaneously present, can cause the pathological phenotype. Therefore, it becomes important in the description of disease pathogenesis to identify as many risk factors for disease prevention and early diagnosis.

DETAILED DESCRIPTION:
Samples collected depending on the disease:

* Peripheral blood;
* Portal blood;
* Saliva;
* Urine;
* Stool;
* Cystic fluid;
* Pancreatic juice;
* Biopsy tissue specimens;

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* signed informed consent

Exclusion Criteria:

* age < 18 years
* unwilling to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biliopancreatic disorders
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of patients with each pancreatic disorder presenting with certain exposures or certain biomarkers | Tthrough study completion, an average of 1 year
  The rate of patients with each pancreatic disorder presenting with certain exposures or certain biomarkers will be evaluated by descriptive statistics and when available compared with that of subjects without such disorders (controls).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Giorgio Arcidiacono, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS OSpedale San Raffaele, Milan, Italy